CLINICAL TRIAL: NCT05827536
Title: Open-label, Randomized, 2-way Crossover, Monocentric, Controlled Study to Evaluate the Effect on Daily PHE Fluctuation of PKU GOLIKE Versus Standard of Care in Patients With Phenylketonuria
Brief Title: Open-label, Randomized, 2-way Crossover, Monocentric, Controlled Study to Evaluate the Effect on Daily PHE Fluctuation of PKU GOLIKE Versus SoC in Patients With PKU.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLK-IT-2023
Record Dates: First submitted 2023-03-24; First posted 2023-04-25 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2023-10

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study products will be self-administered at home according to the assigned randomization sequences, AB or BA where A=standard of care and B=PKU GOLIKE.
  Patients will be randomized in a 1:1 ratio to one of the following two sequences:
  * AB: patients will receive 3 daily self-administrations of their usual standard of care for 2 consecutive days in the first period followed by 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in the second period.
  * BA: patients will receive 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in the first period followed by 3 daily self-administrations of their usual standard of care for 2 consecutive days in the second period. Patients that are not compliant or need to be excluded for other clinical reasons from the treatment schedule will be replaced in order to ensure 20 subjects completing both treatment sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB where A=standard of care and B=PKU GOLIKE (Other): Patients will receive 3 daily self-administrations of their usual standard of care for 2 consecutive days in the first period followed by 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in the second period.
  Interventions: Dietary Supplement: PKU GOLIKE; Dietary Supplement: Standard of Care
- BA where B=PKU GOLIKE and A=standard of care (Other): Patients will receive 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in the first period followed by 3 daily self-administrations of their usual standard of care for 2 consecutive days in the second period.
  Interventions: Dietary Supplement: PKU GOLIKE; Dietary Supplement: Standard of Care

INTERVENTIONS:
Dietary Supplement: PKU GOLIKE — PKU GOLIKE is a food for special medicinal purposes (FSMP) for the dietary management of PKU.
Dietary Supplement: Standard of Care — Protein substitute

SUMMARY:
This is an open-label, randomized, 2-way crossover, monocentric controlled study in patients (≥ 16 years old) with phenylketonuria (PKU).

The comparison will be between the test product (PKU GOLIKE, a prolonged-release amino-acids (AAs) mixture) and standard of care.

DETAILED DESCRIPTION:
The study will consist of a screening visit (V1), two treatment periods with two test days each and a final visit planned at the end of the second treatment period (V2). Test days will occur on two consecutive preferably non-working/school days (T1-T2 and T3-T4,) preferably over two consecutive weeks. Treatment days in the two periods will have to be the same days of the week. T1 should be within two weeks after V1. The study products will be self-administered at home. Following informed consent and verification of eligibility criteria, 20 patients with PKU will be randomized in a 1:1 ratio to one of the following two sequences: AB or BA where A=standard of care and B=PKU GOLIKE. In details:

* AB: patients will receive 3 daily self-administrations of their usual standard of care for 2 consecutive days in the first period followed by 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in thesecond period.
* BA: patients will receive 3 daily self-administrations of PKU GOLIKE for 2 consecutive days in the first period followed by 3 daily self administrations of their usual standard of care for 2 consecutive days in the second period.

No change in the randomization sequence will be allowed.

Each patient will follow the same diet in terms of food, calories and nutrients ranges during the first days (T1 and T3) of each period and the same diet during the second days (T2 and T4) of each period, according to the age and body weight of the patient. The days before the test days each patient will follow her/his standard diet.

PKU GOLIKE /standard of care will be the only protein substitute allowed on each test day, and no sports activities will be allowed on sampling days. Five blood spots will be collected on the second test day of each period. Timing of self-administrations, meals and blood spots will be standardized for each test day. On the test days, no food will be allowed outside of the defined time windows. The first self-administration of each test day will be performed after an overnight fasting (10 -12 h) and before any food intake.

A patient's e-diary will be used to collect information on patient compliance, 24-hour blood spot collections, diet, daily activities, adverse events and event-related concomitant medications.

Adverse events will be continuously monitored during the study, starting from informed consent. Adverse events will be collected by the patients (or by a parent/guardian) in the e-diary and during the telephone calls made by the Investigator to the patients. Moreover, patients (or parents/guardians) will be instructed to promptly report adverse events occurring during the study to the Investigator.

The end of study (V2) will be performed (remotely, by phone) at the end ofthe second treatment period, within 2 weeks after the last test day. Patients prematurely discontinued from the study will be asked to attend (remotely, by phone) a discontinuation visit possibly taking place within 2 weeks from the last test day. At the final/discontinuation visit, the investigator will organize collection of blood spots test and residual PKU GOLIKE product from the patient's domicile through a dedicated courier service. The account of the e-diary will be inactivated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent obtained by the patient prior to beingenrolled into the study and prior to starting any data collection. For legally minor patients, signed written consent shall be obtained also by the parents/legal guardian
2. Male or female, aged ≥16 years.
3. Patients with a registered diagnosis of PKU
4. Ability and willingness to comply with all study procedures and availability for the duration of the study.
5. Patients with mean value of blood Phe >360 µM in the previous 12 months (calculated on at least 3 samples during the previous 12 months; the last sample should be preferably obtained in the 30 days preceding inclusion in the study).
6. Patient taking free-AA and/or GMP as usual amino-acidssupplementation.

Exclusion Criteria:

1. Known or suspected hypersensitivity to any excipients/components of PKU GOLIKE.
2. Treatment with any drug therapy for PKU
3. Patient taking PKU GOLIKE as usual amino-acids supplementation
4. Patient taking LNAA as usual amino-acids supplementation
5. Any moderate to severe medical condition, which in the opinion of the Investigator would interfere with the study procedures or study outcome (reason to be provided)
6. Any current participation in another clinical trial involving investigational or marketed products in the 3 months prior to the inclusion in this study.
7. Pregnancy or lactation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Phe blood concentration with dried blood spots (umol/L) on the second test day with Standard of Care right before product self-administration and before any food intake | at 8:00 am(±15 min) on the second test day with SoC
Phe blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS right before product self-administration and before any food intake | at 8:00 am(±15 min) on the second test day with Golike Plus
Phe blood concentration with dried blood spots (umol/L) on the second test day with Standard of Care right before product self-administration and before food intake | at 12:00 am (±15 min) on the second test day with SoC
Phe blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS right before product self-administration and before food intake | at 12:00 am (±15 min) on the second test day with Golike Plus
Phe blood concentration with dried blood spots (umol/L) on the second test day with Standard of Care before food intake | At 4:00 pm (±15 min) on the second test day with SoC
Phe blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS before food intake | At 4:00 pm (±15 min) on the second test day with Golike Plus
Phe blood concentration with dried blood spots (umol/L) on the second test day with Standard of Care right before product self-administration and before any food intake | at 8:00 pm (±15 min) on the second test day with SoC
Phe blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS right before product self-administration and before any food intake | at 8:00 pm (±15 min) on the second test day with Golike Plus
Phe blood concentration with dried blood spots (umol/L) on the day following the second test day with Standard of Care on the following morning, before any food intake. | at 8:00 am (±15 min) on the day following the second test day with SoC
Phe blood concentration with dried blood spots (umol/L) on the day following the second test day with GOLIKE PLUS on the following morning, before any food intake. | at 8:00 am (±15 min) on the day following the second test day with Golike Plus

SECONDARY OUTCOMES:
Tyr blood concentration with dried blood spots (umol/L) on the second test day with Standard of Care right before product self-administration and before any food intake | at 8:00 am(±15 min) on the second test day with SoC
Tyr blood concentration with dried blood spots (umol/L)on the second test day with GOLIKE PLUS right before product self-administration and before any food intake | at 8:00 am(±15 min)on the second test day with Golike Plus
Tyr blood concentration with dried blood spots (umol/L)on the second test day with Standard of Care right before product self-administration and before any food intake | at 12:00 am(±15 min) on the second test day with SoC
Tyr blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS right before product self-administration and before any food intake | at 12:00 am(±15 min) on the second test day with Golike Plus
Tyr blood concentration with dried blood spots (umol/L)on the second test day with Standard of Care before food intake | at 4:00 pm(±15 min)on the second test day with SoC
Tyr blood concentration with dried blood spots (umol/L) on the second test day with GOLIKE PLUS before food intake | at 4:00 pm(±15 min)on the second test day with Golike Plus
Tyr blood concentration with dried blood spots (umol/L)on the second test day with Standard of Care right before product self-administration and before any food intake | at 8:00 pm(±15 min) on the second test day with SoC
Tyr blood concentration with dried blood spots (umol/L)on the second test day with GOLIKE PLUS right before product self-administration and before any food intake | at 8:00 pm(±15 min) on the second test day with Golike Plus
Tyr blood concentration with dried blood spots (umol/L)on the day following the second test day with Standard of Care on the following morning, before any food intake. | at 8:00 am(±15 min) on the day following the second test day with SoC
Tyr blood concentration with dried blood spots (umol/L) on the day following the second test day with GOLIKE PLUS on the following morning, before any food intake. | at 8:00 am(±15 min) on the day following the second test day with Golike Plus

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Rovelli, MD, Principal Investigator — ASST Santi Paolo e Carlo, Presidio Ospedale San Paolo, Via Antonio di Rudinì 8 - 20142, Milano (Italy)
Locations (1):
- ASST Santi Paolo e Carlo, Presidio Ospedale San Paolo, Via Antonio di Rudinì 8, Milan, Italy